CLINICAL TRIAL: NCT05770934
Title: The Effectiveness of Late-initiated Blood Flow Restricted Rehabilitation Exercises on Functional Capacity, Lower Limb Muscle Strength and Patient-reported Outcomes After Total Knee Replacement
Brief Title: Late-initiated Blood Flow Restricted Rehabilitation Exercises After Total Knee Replacement
Acronym: EXKnee2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No participant wanted to participate
Sponsor: University of Aarhus (Other)
Collaborators: Horsens Hospital (Other); Regionshospitalet Silkeborg (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXKnee late phase
Record Dates: First submitted 2021-06-24; First posted 2023-03-16 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis, Knee; Arthropathy of Knee
Keywords: Rehabilitation; Blood flow restriction exercise; Total knee replacement; Functional Capacity
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- home-based BFRE (Experimental): Patients in the home-based BFRE group will be carefully instructed in how to perform the exercise program with four weekly sessions for 12 weeks (48 training sessions within an 84-day period). Each session will consist of one lower-limb resistance training exercise: sit-to-stand from a ~43 cm high chair. The exercise will consist of four rounds interspaced by a 30-seconds rest pause. The first, second, and third round will consist of 30, 15, 15 repetitions, while the fourth round will be performed until volitional fatigue. The patients will be instructed to perform both the eccentric and concentric contractions at a steady 2-sec pace with, preferably, no time for relaxation in the transition from eccentric to concentric phase (i.e. the bottom is only "kissing" the chair before reversing the movement upwards). When a patient can perform more than 25 repetitions in the last round, they are encouraged to add external resistance corresponding to around 5 kg.
  Interventions: Other: Blood flow restricted low-load resistance exercise
- Control Group (No Intervention): Patients in the control group will performed the same tests 12 months after surgery and 15 months after surgery as the intervention home-based BFRE group.

INTERVENTIONS:
Other: Blood flow restricted low-load resistance exercise — Blood flow restricted low-load resistance exercise
  Arms: home-based BFRE

SUMMARY:
This trial will investigate the effectiveness of applying low-load blood flow restricted exercise 12 months after receiving a total knee replacement to achieve a functional capacity-level similar to healthy peers. Participants will be allocated to either an exercise group performing a sit-to-stand exercise 4/weekly with concurrent partial restriction of the blood flow to the limbs or a usual care.

DETAILED DESCRIPTION:
Blood flow restricted exercise (BFRE) is resistance training with low loads (30% 1repetition maximum (RM) performed with concurrent partial blood flow restriction by means of pneumatic cuff compression around the working limb.

Group 1:

BFRE group: After being introduced to the exercise principles, the participants will perform 4/weekly home-based BFRE sessions for 12 weeks from. Each session will consist of a sit-to-stand exercise performed with concurrent partial restriction of the blood flow to the limbs. The exercise consist of 4 rounds interspaced by 30 seconds of rest. 1st round: 30 repetitions (reps); 2nd round: 15 reps; 3rd round: 15 reps; 4th round: until exhaustion. Patients will rest in a standardized resting position between each set to maintain the desired resting cuff-pressure.

The occlusion pressure will be set at 60% of total limb occlusion pressure and starting load intensity will be 30% 1repetition maximum (1RM) in both exercises. If patients can perform more than 15 repetitions in the 4th exercise set, more external resistance will added at the next session.

Group 2:

CON group: Will follow standard procedures 12 months after total knee replacement.

The trial is designed as a multicenter (two sites) randomized controlled trial. The primary outcome, Timed Up and Go, as well as all secondary outcomes measured at end of intervention.

The patients in the present project will be recruited from the patients in Jorgensen et al. (1) who have either performed 8 weeks of preoperative BFRE (PREBFR), received usual care prior to total knee replacement (TKR) (PRECON), or participated in the cohort-study. Further, exclusion criteria will remain the same as in Jorgensen et al. (1).

before, enrollment all patients will be re-screened for eligibility by the principal author (SLJ) who will perform the inclusion of patients and provide oral and written project information. All patients accepting to participate will sign a written informed consent to participate in the project. All patients who have participated in the randomized controlled trial will be offered 12 weeks of home based BFRE, while all subject who have participated in the cohort-study will be invited to serve as a control group

Patients in the home based BFRE group will be carefully instructed in how to perform the BFRE exercises at home.

The aim of the current study is to investigate the effectiveness of 12 weeks of BFRE homed-based exercises initiated 12 months after TKR. Furthermore, we will determine if patients who have performed 8 weeks of preoperative BFRE profits more from the late initiated BFRE program compared to patients who have not received 8 weeks of preoperative BFRE.

All descriptive statistics and tests will be reported in accordance with the recommendations of the "Enhancing the QUAlity and Transparency Of health Research" (EQUATOR) network and the CONSORT statement. Intention-to-treat principle (i.e. all patients as randomized independent of departures from allocation treatment, compliance and/or withdrawals) and per protocol analysis will be conducted. A one-way analysis of variance (one-way ANOVA) model will be used to analyze between mean change in continuous outcome measures between the group of patients who have performed 8 weeks of preoperative BFRE (PREBFR) and the group who did not perform 8 weeks of preoperative BFRE (PRECON) (27). The model includes changes from baseline to end of intervention. Also, to gain insight into the potential pre-to-post training differences within the whole patient population (PREBFR+PROCON), the PREBFR-patients and the PRECON-participants, paired student t-tests will be performed. Level of statistical significance is P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the EXknee project (Efficacy of low-load blood flow restricted resistance EXercise in patients with Knee osteoarthritis scheduled for total knee replacement (EXKnee) Jorgensen et al. 2020)

Exclusion Criteria:

* Severe cardiovascular diseases (New York Heart Association class III and IIII), -
* previous stroke incident, thrombosis incident
* Traumatic nerve injury in affected limb
* Unregulated hypertension (Systolic ≥180 or diastolic ≥110 mmHg)
* Spinal cord injury
* Cancer diagnosis and currently undergoing chemo-, immuno-, or radiotherapy
* Inadequacy in written and spoken Danish
* living more than 45 minutes from either Horsens Regional Hospital or Silkeborg Regional Hospital.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
30-seconds chair stand test (30-CST) | 1 year after surgery
  The 30s-CST measures the number of sit-to-stand repetitions completed within 30 seconds. Patients will be instructed to perform a sit-to-stand movement starting from a seated position (seat height 43 cm without armrests) having the feet placed flat on the floor shoulder width apart, and arms crossed on chest to a standing position (hip and knee joints fully extended) repeated as many times as possible for 30 seconds
Change in 30-seconds chair stand test (30-CST) | 15 months after surgery
  The 30s-CST measures the number of sit-to-stand repetitions completed within 30 seconds. Patients will be instructed to perform a sit-to-stand movement starting from a seated position (seat height 43 cm without armrests) having the feet placed flat on the floor shoulder width apart, and arms crossed on chest to a standing position (hip and knee joints fully extended) repeated as many times as possible for 30 seconds

SECONDARY OUTCOMES:
Timed Up & Go (TUG) | 1 yeay after surgery
  The TUG assesses the time required for patients to stand from a chair (seat height 46 cm) walk around a tape mark 3 meters away and sit into the chair at return.
Timed Up & Go (TUG) | 15 months after surgery
  The TUG assesses the time required for patients to stand from a chair (seat height 46 cm) walk around a tape mark 3 meters away and sit into the chair at return.
4x10 meter fast-paced walk test (40m-FWT) | 1 year after surgery
  The 40m fast-paced walk test (40m-FWT) measures the total time taken to walk 4 x 10 m excluding turns (meter/sec).
4x10 meter fast-paced walk test (40m-FWT) | 15 months after surgery
  The 40m fast-paced walk test (40m-FWT) measures the total time taken to walk 4 x 10 m excluding turns (meter/sec).
Isometric knee extensor strength | 1 year after surgery
  Isometric knee extensor muscle strength will be measured with the participants seated on a examination table with knees and hip positioned at 90 degree flexion. Assessment of muscle strength will be performed with a hand-held dynamometer, fixed with an adjustable rigid belt to the examination table.
Isometric knee extensor strength | 15 months after surgery
  Isometric knee extensor muscle strength will be measured with the participants seated on a examination table with knees and hip positioned at 90 degree flexion. Assessment of muscle strength will be performed with a hand-held dynamometer, fixed with an adjustable rigid belt to the examination table.
Isometric knee flexor strength | 1 year after surgerty
  Isometric knee flexor muscle strength will be measured with the participants seated on a examination table with knees and hip positioned at 90 degree flexion. Assessment of muscle strength will be performed with a hand-held dynamometer, fixed with an adjustable rigid belt to the examination table
Isometric knee flexor strength | 15 months after surgery
  Isometric knee flexor muscle strength will be measured with the participants seated on a examination table with knees and hip positioned at 90 degree flexion. Assessment of muscle strength will be performed with a hand-held dynamometer, fixed with an adjustable rigid belt to the examination table
Knee disability and Osteoarthritis Outcome Score (KOOS) | 1 year after surgery
  KOOS is a patient-administered knee specific questionnaire comprising five subscales Pain; Symptoms; Activities of daily living; Sport & Recreation; and Knee-Related Quality of Life.
Knee disability and Osteoarthritis Outcome Score (KOOS) | 15 months after surgery
  KOOS is a patient-administered knee specific questionnaire comprising five subscales Pain; Symptoms; Activities of daily living; Sport & Recreation; and Knee-Related Quality of Life.
EuroQol Group 5-dimension (EQ-5D-5L)after surgery | 1 year after surgery
  The EQ-5D-L5 is a self-completion questionnaire consisting of two parts; first part of the EQ-5D-5L comprises five dimensions involving mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
EuroQol Group 5-dimension (EQ-5D-5L)after surgery | 15 months after surgery
  The EQ-5D-L5 is a self-completion questionnaire consisting of two parts; first part of the EQ-5D-5L comprises five dimensions involving mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Adverse events | 15 months after surgery
  Adverse events will be defined as unpredicted or unintended events, signs, or disease occurring during the period from inclusion until follow-up resulting in contact with the healthcare system (hospital or general practitioner) independent of whether or not the event is related to the intervention or outcome assessments
Exercise compliance and progression | 15 months after surgery
  The participants will report their adherence, experience and understanding of the training in a training diary
Numeric Rating Scale Pain (NRS pain) | 1 year after surgery
  The NRS for pain is a segmented unidimensional 11-item measure of pain intensity in adults
Numeric Rating Scale Pain (NRS pain) | 15 months after surgery
  The NRS for pain is a segmented unidimensional 11-item measure of pain intensity in adults
Numeric Rating Scale Pain (NRS pain) | during 12 weeks exercise program
  The NRS for pain is a segmented unidimensional 11-item measure of pain intensity in adults

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Hospital Horsens, Horsens, Horsens, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Regional Hospital Horsens is responsible for handling all personal data provided by both sites in accordance to the Clinical Trial Agreement and the EU General Data Protection Regulation (GDPR)